CLINICAL TRIAL: NCT06956586
Title: The Ethical Approval From Gazi University Has Been Obtained.The Institutional Approval From Bilkent City Hospital Has Been Obtained.
Brief Title: Therapeutic Communication Techniques for Children Aged 7-12 in Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Özge Köksal, Child Health and Disease Nursing Department Research Assistant, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-14774941-199-996608
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Emotional States; Therapeutic Communication in Pediatric ICU; Child Emotional Well-being in ICU
Keywords: Therapeutic Communication; Intensive Care Unit (ICU); Pediatric Care; Child Psychological Support

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Communication Techniques (Experimental): Participants in the intervention group will participate in therapeutic communication sessions using storytelling and drawing techniques for 2 days.
  Interventions: Other: Therapeutic communication techniques
- Standard Care (No Intervention): The control group will receive standard care. After the study is completed, therapeutic communication techniques will also be applied to the control group

INTERVENTIONS:
Other: Therapeutic communication techniques — Therapeutic communication techniques will be applied to children in the intensive care unit for two days."
  Arms: Therapeutic Communication Techniques

SUMMARY:
Summary of the Research Children may need to stay in intensive care for a period of time due to acute or chronic illnesses in their lives.There may be anxiety, fear and concerns in intensive care. Therefore, a healthy communication with the child, such as care, accurate transfer and reporting of the events and situations experienced according to the development level, the use of appropriate therapeutic communication, the child's mental and spiritual life includes all lives. The aim of this study is to examine the effects of therapeutic communication techniques applied to the 7-12 age groups in intensive care on the emotional development of children. The research will be patterned later. The research storage will consist of 70 children between the ages of 7-12 who are hospitalized in the Intensive Care Unit of Ankara Bilkent City Hospital Pediatric Intensive Care Unit and Uşak University Education and Research Hospital. Data will be collected with 1. Descriptive Data Form Related to the Child and Family, 2. State Anxiety Inventory, 3. Koppitz's Human Figure Drawing Test, 4. "Facial Expressions Rating Scale" in Wong and Baker.

Purpose of the study: The purpose of this study is to examine the effects of therapeutic communication techniques applied to children aged 7-12 in intensive care on the emotional state of the children.

Hypotheses of the Study:

H1.1: The average total score of the state anxiety scale in the intervention group (children receiving therapeutic communication techniques) will differ from that of the control group (children not receiving therapeutic communication techniques).

H1.2: The emotional state of the children in the intervention group, as measured by the Koppitz Human Figure Drawing Test, will differ from the emotional state of children in the control group.

Before the therapeutic communication method is applied to the children in the intervention and control groups, the descriptive characteristics data form, the State Anxiety Inventory, the Facial Expressions Rating Scale, and the Emotion Wheel will be applied.

The forms will be shown to the child by the researcher at the child's bedside in the intensive care unit and filled out face to face by the researcher. After the therapeutic communication intervention is completed, Koppitz's Human Figure Drawing Test and State Anxiety Inventory will be applied to the children in the intervention and control groups. The estimated application time of the forms is 30 minutes. The application will last 2 days.

DAY 1: Application of joint storytelling as a therapeutic communication technique by the researcher to the children DAY 2: Application of picture drawing technique as a therapeutic communication technique by the researcher to the children

DETAILED DESCRIPTION:
Study Design: study is designed as a randomized controlled trial to evaluate the effects of therapeutic communication techniques on the emotional development of children aged 7-12 in intensive care units.

Participants:

The study will include 70 children aged 7-12 years who are admitted to the Pediatric Intensive Care Units of Ankara Bilkent City Hospital and Uşak University Training and Research Hospital.

Randomization:To reduce selection bias and control for variables that may affect outcome parameters, participants will be randomly assigned to either the intervention group, which will receive therapeutic communication techniques, or the control group, which will receive standard care.In order to ensure homogeneity between groups, it will be created with the existing stratification method.The CONSORT 2022 (Updated Guidelines for Reporting Randomized Parallel Group Trials) report will be followed during the randomization phase The data obtained in the study will be evaluated in the computer environment with the SPSS 27.0 package data program. The conformity of the data to normal distribution will be examined with descriptive statistics (skewness, kurtosis), hypothesis tests (Kolmogorov-Smirnov/Shapiro-Wilk tests) and visually (histogram and probability graphs). In comparisons between groups, single-factor covariance analysis (ANCOVA) will be applied to eliminate bias in normally distributed data, and Mann Whitney U test will be applied for non-normally distributed data. In intra-group evaluations, the significance test of the difference between two pairs will be used for normally distributed ordinal data, and the Wilcoxon paired two-sample test will be used for non-normally distributed ones. Chi-square test will be used in comparisons of nominal data between groups.

Ethical Aspects of the Research A permit numbered 09 dated 12.07.2024 was obtained from the Gazi University Ethics Committee for the implementation of the data collection forms. Written consent will be obtained from the patient child and his/her family to be included in the study, and the identity and medical conditions of the participants will be kept confidential. The children in the control group will be subjected to the technique of drawing pictures and telling stories after the study.

ELIGIBILITY:
Inclusion Criteria

Aged between 7 and 12 years,

Receiving treatment in an intensive care unit,

Children and families who agree to participate in the study,

Conscious with a Glasgow Coma Scale (GCS) score of 15,

First-time experience in an intensive care unit,

Able to speak and understand Turkish,

Not experiencing intense symptoms such as pain or nausea during the procedure,

Children monitored at levels 1 and 2 will be included.

Exclusion Criteria

The child has a chronic illness requiring frequent hospitalizations and treatment,

The child has a medically diagnosed psychological disorder.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | Before and immediately after the application of therapeutic communication techniques."
  The State-Trait Anxiety Inventory is a psychological inventory that measures the level of anxiety in individuals. It consists of two separate scales: one that measures state anxiety (the temporary anxiety experienced at a specific moment or situation) and one that measures trait anxiety (the general tendency to experience anxiety in a variety of situations).It was developed to assess how children feel at that moment. It consists of 20 items and aims to assess feelings related to state anxiety. The options in this form are scored as "not at all" (1), "a little" (2), "a lot" (3), "always" (4). The highest score that can be obtained from the State Anxiety Inventory is 80 and the lowest score is 20. A high score indicates a high anxiety state. A low score indicates a low anxiety state.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Emeksiz, Assoc. Prof., Study Director — Bilkent City Hospital; Ebru Kılıçarslan, Professor, Study Director — Gazi Univercıty; Özge Köksal, Research Assistant, Principal Investigator — Uşak Univercıty
Locations (1):
- Ankara Bilkent City Hospital, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rennick JE, Stremler R, Horwood L, Aita M, Lavoie T, Majnemer A, Antonacci M, Knox A, Constantin E. A Pilot Randomized Controlled Trial of an Intervention to Promote Psychological Well-Being in Critically Ill Children: Soothing Through Touch, Reading, and Music. Pediatr Crit Care Med. 2018 Jul;19(7):e358-e366. doi: 10.1097/PCC.0000000000001556. PMID 29659416
- [Derived] Koksal O, Kilicarslan E, Emeksiz S. Drawing and mutual storytelling to alleviate anxiety and improve emotional well-being in children in PICU: a randomized controlled trial. Eur J Pediatr. 2025 Sep 5;184(9):602. doi: 10.1007/s00431-025-06454-5. PMID 40913193
- See also: Ankara Bilkent City Hospital — https://ankarasehir.saglik.gov.tr/
- Available data/document: Study Protocol: Research — https://pubmed.ncbi.nlm.nih.gov/37330438/ — There is no additional information."